CLINICAL TRIAL: NCT03886428
Title: Lunch Feeding Study for Men and Women
Brief Title: The Influence of Satiation Measures on the Portion Size Effect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Jenny Craig, Inc. (Industry)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutrition and Director of the Laboratory for the Study of Human Ingestive Behavior, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PortionSize106
Record Dates: First submitted 2019-03-14; First posted 2019-03-22 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Feeding Behavior
MeSH Terms: conditions — Feeding Behavior | interventions — Portion Size

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 100% Portion Size (Experimental): Test meal with portion size 100% of baseline
  Interventions: Other: 100% portion size
- 125% Portion Size (Experimental): Test meal with portion size 125% of baseline
  Interventions: Other: 125% portion size
- 150% Portion Size (Experimental): Test meal with portion size 150% of baseline
  Interventions: Other: 150% portion size
- 175% Portion Size (Experimental): Test meal with portion size 175% of baseline
  Interventions: Other: 175% portion size

INTERVENTIONS:
Other: 100% portion size — Entree portion size 100% of baseline
  Arms: 100% Portion Size
Other: 125% portion size — Entree portion size 125% of baseline
  Arms: 125% Portion Size
Other: 150% portion size — Entree portion size 150% of baseline
  Arms: 150% Portion Size
Other: 175% portion size — Entree portion size 175% of baseline
  Arms: 175% Portion Size

SUMMARY:
The purpose of this study is to gain a better understanding of the satiation measures that influence human eating behavior in regard to intake of large portion sizes at a meal. The investigators hypothesize that satiation measures will influence the magnitude of the portion size effect at a meal. Additionally, other individual characteristics will be examined for their influence on the portion size effect. The portion size effect will be measured by serving a test meal once a week for four weeks in which the portion size of the entree will be varied.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to travel to Penn State University Park campus weekly for meals
* Be a man or woman 18 - 70 years old
* Regularly eat 3 meals/day
* Be willing to avoid alcohol the day before and during test days
* Have a body mass index between 18.0 and 35.0 kg/m*m
* Be willing to refrain from eating after 10 pm the evening before test sessions
* Be willing to participate in all study procedures

Exclusion Criteria:

* Must not be a smoker
* Must not be an athlete in training
* Must not be pregnant or breastfeeding at the time of screening
* Have taken prescription or non-prescription drugs that may affect appetite or food intake within the last 3 months
* Dislike or be unable to eat the test foods (because of allergies, intolerance, or dietary restrictions)
* Must not be currently dieting to gain or lose weight
* Have a health condition that affects appetite
* Have participated in a similar study in our lab in the past year
* Must not be a student, faculty, or staff member in nutritional sciences or psychology

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Change in energy intake | Weeks 1, 2, 3, 4
  Calculated energy intake (kcal) based on weight and energy density of food consumed
Change in intake by weight | Weeks 1, 2, 3, 4
  Weights (grams) of all foods consumed

SECONDARY OUTCOMES:
Change in bite count | Weeks 1, 2, 3, 4
  The number of bites of the entree during the meal
Change in meal duration | Weeks 1, 2, 3, 4
  Duration of the meal in seconds
Change in mean bite rate | Weeks 1, 2, 3, 4
  Assessed from meal duration (seconds) and number of bites taken
Change in mean bite size | Weeks 1, 2, 3, 4
  Assessed from entree intake (grams) and number of bites
Change in mean eating rate | Weeks 1, 2, 3, 4
  Assessed from entree intake (grams) and meal duration
Change in distribution of estimated bite size | Weeks 1, 2, 3, 4
  Assessed as small or large bites from video observation
Change in sip count | Weeks 1, 2, 3, 4
  The number of sips of the water during the meal
Change in rating of the pleasantness of the taste of the entree sample | From before the test meal to after the test meal in weeks 1, 2, 3, 4
  Measured on a 100-mm visual analogue scale ranging from not at all pleasant (0 mm) to extremely pleasant (100 mm). This will be used to calculate Sensory-Specific Satiety
Change in rating of the pleasantness of the taste of food samples | From before the test meal to after the test meal in weeks 1, 2, 3, 4
  Measured on a 100-mm visual analogue scale ranging from not at all pleasant (0 mm) to extremely pleasant (100 mm). This will be used to calculate Sensory-Specific Satiety
Change in rating of prospective consumption of the entree sample | From before the test meal to after the test meal in weeks 1, 2, 3, 4
  Measured on a 100-mm visual analogue scale ranging from none at all (0 mm) to vary large amount (100 mm) in answer to the question 'How much of the pasta do you want to eat right now?'. This will be used to calculate Sensory-Specific Satiety
Change in rating of prospective consumption of food samples | From before the test meal to after the test meal in weeks 1, 2, 3, 4
  Measured on a 100-mm visual analogue scale ranging from none at all (0 mm) to vary large amount (100 mm) how much of the [this food] do you want to eat right now?. This will be used to calculate Sensory-Specific Satiety
Change in rating of hunger | From before the test meal to after the test meal in weeks 1, 2, 3, 4
  Measured on a 100-mm visual analogue scale ranging from not at all hungry (0 mm) to extremely hungry (100 mm)
Change in rating of thirst | From before the test meal to after the test meal in weeks 1, 2, 3, 4
  Measured on a 100-mm visual analogue scale ranging from not at all thirsty (0 mm) to extremely thirsty (100 mm)
Change in ratings of prospective consumption | From before the test meal to after the test meal in weeks 1, 2, 3, 4
  Measured on a 100-mm visual analogue scale ranging from nothing at all (0 mm) to a large amount (100 mm) in answer to the question 'How much food could you eat right now?'.
Change in ratings of nausea | From before the test meal to after the test meal in weeks 1, 2, 3, 4
  Measured on a 100-mm visual analogue scale ranging from not at all nauseated (0 mm) to extremely nauseated (100 mm)
Change in rating of fullness | From before the test meal to after the test meal in weeks 1, 2, 3, 4
  Measured on a 100-mm visual analogue scale ranging from not at all full (0 mm) to extremely full (100 mm)

OTHER OUTCOMES:
Rating of the size of the entree compared to participants' usual portion | At the start of the test meal in weeks 1, 2, 3, 4
  100-point visual analog scale ranging from a lot smaller to a lot larger
Rating of how filling participants expect this amount of food to be | At the start of the test meal in weeks 1, 2, 3, 4
  100-point visual analog scale ranging from not at all filling to extremely filling
Rating of pleasantness of taste of entree | At the start of the test meal in weeks 1, 2, 3, 4
  100-point visual analog scale ranging from not pleasant at all to extremely pleasant
Ratings of Meal Termination due to fullness | At the end of the test meal in weeks 1, 2, 3, 4
  100-point visual analog scale ranging from strongly disagree to strongly agree
Ratings of Meal Termination due to eating their usual amount | At the end of the test meal in weeks 1, 2, 3, 4
  100-point visual analog scale ranging from strongly disagree to strongly agree
Ratings of Meal Termination due to eating is no longer a priority | At the end of the test meal in weeks 1, 2, 3, 4
  100-point visual analog scale ranging from strongly disagree to strongly agree
Ratings of Meal Termination due to there being no food left | At the end of the test meal in weeks 1, 2, 3, 4
  100-point visual analog scale ranging from strongly disagree to strongly agree
Ratings of Meal Termination due to self-consciousness about amount consumed | At the end of the test meal in weeks 1, 2, 3, 4
  100-point visual analog scale ranging from strongly disagree to strongly agree
Ratings of Meal Termination due to the food no longer tasting good | At the end of the test meal in weeks 1, 2, 3, 4
  100-point visual analog scale ranging from strongly disagree to strongly agree
Rating of proportion of meal eaten | At the end of the test meal in weeks 1, 2, 3, 4
  100-point visual analog scale ranging from 0% to 100%
Rating of calories consumed at the meal | At the end of the test meal in weeks 1, 2, 3, 4
  Open ended question

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No